CLINICAL TRIAL: NCT05387824
Title: Comparison of the Efficacy of Transcutaneous Tibial Nerve Stimulation and Extracorporeal Magnetic Stimulation in Women With Idiopathic Overactive Bladder
Brief Title: Tibial Nerve and Extracorporeal Magnetic Stimulation for Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Medical Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sn 60116787-020/59365
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Idiopathic Overactive Bladder; Bladder Training; Transcutaneous Tibial Nerve Stimulation; Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Bladder Training - Control group (Active Comparator): BT, consisting of four stages, won't contain any PFMT programs in all groups. In these stages, including urgency supression strategies, it was aimed to delay urination, to inhibit detrusor contraction and to prevent urgency; by squeezing the PFM several times in a row (women will be encouraged to pause/ stop their work, sit down if possible, relax the entire body and squeeze PFM repeatedly), breathing deeply, giving their attention to another job for a while and self-motivating (I can do it, I can check the urination, etc.).
  Interventions: Behavioral: Bladder Training
- Group 2: Bladder Training + TTNS (Experimental): Two self-adhesive surface electrodes will be positioned according to the protocol which previously explained, with the negative electrode 2 cm behind the medial malleolus and positive electrode 10 cm proximal. Correct positioning wil be determined by noting a hallux reaction (plantar flexion of great toe or fanning of all toes). The stimulation protocol will be delivered at fixed 20 Hz and pulse width 200 ms in continous mode in accordance with the PTNS stimulation protocol. The intensity of the stimulation current (range 0-50 mA) will be determined once correct positioning are established, according to the comfort level of the person. TTNS sessions will be performed twice a week for 6 weeks. Every session will be lasted 30 min. Treatment will consist of 12 sessions of stimulation.
  Interventions: Device: Electrical Stimulation- TTNS; Behavioral: Bladder Training
- Group 3: Bladder Training + MStim (Experimental): Patients are told to sit on the chair with a magnetic coil below the chair. When a volume conductor is in serted by this magnetic field, an eddy current flow is generated. This eddy current stimulates nerve or muscle of the pelvic floor. To apply MS, the device will be set to generate its maximum stimuli, with a stimulation pulse width of 200 μs and a stimulation repetition cycle of 10 Hz in accordance with the literature. When setting the device at each treatment session, patients will be interviewed so that they receive the stimuli at the maximum stimulation intensity (maximum tolerable stimulation intensity) .
  Interventions: Device: Magnetic stimulation -Armchair type MS • NovaMag NT-60; Behavioral: Bladder Training

INTERVENTIONS:
Device: Magnetic stimulation -Armchair type MS • NovaMag NT-60 — MS was applied two days a week, 20 minutes a day, a total of 12 sessions for 6 weeks.
  Arms: Group 3: Bladder Training + MStim
Device: Electrical Stimulation- TTNS — TTNS were performed 2 days a week, for 30 min a day, for a total of 12 sessions for 6 weeks.
  Arms: Group 2: Bladder Training + TTNS
Behavioral: Bladder Training — Control group All women were informed about BT for 30 minutes. Then it was given as a written brochure to be implemented as a home program.
  BT, consisting of four stages, did not contain any PFMT programs in two groups.

SUMMARY:
Overactive bladder (OAB) syndrome is urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of urinary tract infection. For the treatment of OAB; pharmacological and non-pharmacological methods are available. The availability and the continuation rate of pharmacological treatments are lower than non-pharmacological treatments due to side effects.

Non-pharmacologic treatment methods are evaluated in two groups as active and passive methods. Active methods which active participation of the patient is required during treatment are Pelvic floor muscle exercise (PFME), biofeedback assisted PFME, vaginal cones, while passive methods are Electrical Stimulation, extracorporeal Magnetic Stimulation (MStim) and Transcutaneous Tibial Nerve Stimulation (TTNS) techniques.

In this study, investigators aim to evaluate the effectiveness of TTNS and extracorporeal MStim, which are noninvasive methods, added to bladder training (BT) in women with OAB, with a prospective randomized controlled research method.

DETAILED DESCRIPTION:
This study is a prospectively randomized, controlled trial. The trial will be held at Urogynecological Rehabilitation Unit of Pamukkale University, Physical Medicine and Rehabilitation Department between Nisan 2022 and October 2022. The local ethics committee approved the study (approvel no: 60116787-020/59365).

Participants will be informed about the purpose and contents of the study and all women give written consent to participate. By using a random number generator, all participants who include the study will be randomized into three groups as follows: The Group 1 will receive BT program alone, the Group 2 will be applied to BT plus TTNS, The Group 3 was applied to BT plus MStim.

Group 1: BT - Control group:

All women will be informed about BT for 30 minutes. Then it will be given as a written brochure to be implemented as a home program.

BT, consisting of four stages, will not contain any PFMT programs in anyone of three groups.

Group 2: BT plus TTNS:

Two self-adhesive surface electrodes will be positioned according to the protocol previously used with the negative electrode 2 cm behind the medial malleolus and positive electrode 10 cm proximal. Correct positioning will be determined by noting a hallux reaction (plantar flexion of great toe or fanning of all toes). The stimulation protocol will be delivered at fixed 20 Hz and pulse width 200 ms in continous mode in accordance with the PTNS stimulation protocol. The intensity of the stimulation current (range 0-50 mA) will be determined once correct positioning was established, according to the comfort level of the person. TTNS sessions will be performed twice a week for 6 weeks. Every session will be lasted 30 min. Treatment will consist of 12 sessions of stimulation.

Group 3: BT plus MStim:

Pariticipants will be told to sit on the chair with a magnetic coil below the chair. When a volume conductor is in serted by this magnetic field, an eddy current flow is generated. This eddy current stimulates nerve or muscle of the pelvic floor. To apply MStim, the device will be set to generate its maximum stimuli, with a stimulation pulse width of 200 μs and a stimulation repetition cycle of 10 Hz in accordance with the literature (10,13-15). When setting the device at each treatment session, participants will be interviewed so that they'll receive stimuli at the maximum stimulation intensity (maximum tolerable stimulation intensity). MStim will be applied two days a week, 20 minutes a day, a total of 12 sessions for 6 weeks. MStim sessions will be performed by other physician.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with clinical diagnosis of idiopathic OAB Urodynamically confirmed detrusor overactivity (the presence of detrusor contractions in the filling phase of saline cystometry)
* Not tolerated or unresponsive to antimuscarinics and discontinued at least 4 weeks Able to give written, informed consent Able to understand the precedures, advantages and possible side effects Willing and able to complate the voiding diary and QoL questionnaire The strength of PFM 3/5 and more

Exclusion Criteria:

* History of BT, MS therapy
* Pregnancy or intention to become pregnant during the study Current vulvovaginitis or urinary tract infections or malignancy
* More than stage 2 according to the pelvic organ prolapse quantification (POP-Q)
* Cardiac pacemaker, implanted defibrillator, coronary artery stent
* Ongoing treatment for arrhythmia
* Lower abdominal pain or dysmenorrhea
* yet to be diagnosed Electronic device or metallic implant applied to areas between the lumbar region and lower extremities
* Previous urogyneceological surgery within 3 months
* Ongoing surgical treatment or treatment with implantable devices for urinary incontinence or use of intrauterin copper devices
* Neurogenic bladder, signs of neurologic abnormalities at objective examination; history of the peripheral or central neurologic pathology
* Ultrasonographic evidence of PVR volume more than 100 ml

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women over the age of 18 with clinical diagnosis of idiopathic OAB and urodynamically confirmed detrusor overactivity (the presence of detrusor contractions in the filling phase of saline cystometry).
Enrollment: 66 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Incontinence episodes | 6 weeks
  Patients with a 50% or greater reduction in incontinence episodes were consider positive responders

SECONDARY OUTCOMES:
Severity of incontinence | 6 weeks
  The 24-hour pad test was carried out to evaluate urinary loss.
Nocturia | 6 weeks
  It was used "nocturia" from data collected with a 3-day bladder diary.
Frequency | 6 weeks
  It was used "frequency" from data collected with a 3-day bladder diary.
Number of pads | 6 weeks
  It was used "number of pads" from data collected with a 3-day bladder diary.
Symptom severity | 6 weeks
  Overactive Bladder Questionnaire (OAB-V8) was used to evaluate symptom severity in patients with in the study. Minimum score is 0, maximum score is 40 and high scores mention worse outcome.
QoL | 6 weeks
  The Incontinence Impact Questionnaire (IIQ-7) scale which has great validity in studies was used to assess the patient's QoL associated with incontinence problem. Minimum score is 0, maximum score is 21 and high scores mention worse outcome.
improvement rate | 6 weeks
  The improvement was assessed in terms of 50% and more reduction in wet weight compared to baseline measurements in the 24-hour pad test.
24-hour pad test (Cure) | 6 weeks
  In 24-hour pad test, 1.3 gr under of it was considered as a cure.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz N, Oztekin SNS, Akkoc Y. Comparison of Magnetic and Transcutaenous Tibial Nerve Stimulation Added to Bladder Training for Overactive Bladder: A Randomized Controlled Trial. Int Urogynecol J. 2025 Dec;36(12):2379-2388. doi: 10.1007/s00192-025-06215-w. Epub 2025 Jul 7. PMID 40622410